CLINICAL TRIAL: NCT05150041
Title: A Pilot Study for the Efficacy of Guardian Connect to Modify Lifestyle in Patients With Type 2 Diabetes Mellitus
Brief Title: The Efficacy of Guardian Connect to Modify Lifestyle in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Cheol-Young Park, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KBSMC 2019-04-021
Record Dates: First submitted 2019-10-09; First posted 2021-12-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes self-management education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iPRo2 only (Control group) (Active Comparator): - The Control group will go through target lifestyle coaching including diet and exercise and they will undergo 24 weeks of follow-up period.
  Interventions: Device: iPro2
- iPRo2 + RT-CGM 1 week treatment (Treatment group 1) (Experimental): Treatment group 1 will go through target lifestyle coaching including diet and exercise and will have 1 session of RT-CGM after which they will undergo 24 weeks of follow-up period.
  Interventions: Device: Guardian connect; Device: iPro2
- iPRo2 + RT-CGM 1 week on /3 weeks off (2cycles) (Treatment 2) (Experimental): - Treatment group 2 will go through target life coaching including diet and exercise and will have 2 sessions(CGM 1week, 12week after measuring HbA1c) of RT-CGM after which they will undergo 24 weeks of follow-up period.
  Interventions: Device: Guardian connect; Device: iPro2

INTERVENTIONS:
Device: Guardian connect — * Treatment group 1 will go through target lifestyle coaching including diet and exercise and will have 1 session of RT-CGM after which they will undergo 24 weeks of follow-up period.
  * Treatment group 2 will go through target life coaching including diet and exercise and will have 2 sessions(CGM 1week, 12week after measuring HbA1c) of RT-CGM after which they will undergo 24 weeks of follow-up period.
  Arms: iPRo2 + RT-CGM 1 week on /3 weeks off (2cycles) (Treatment 2); iPRo2 + RT-CGM 1 week treatment (Treatment group 1)
Device: iPro2 — * Treatment group 1 will go through target lifestyle coaching including diet and exercise and will have 1 session of RT-CGM after which they will undergo 24 weeks of follow-up period.
  * Treatment group 2 will go through target life coaching including diet and exercise and will have 2 sessions(CGM 1week, 12week after measuring HbA1c) of RT-CGM after which they will undergo 24 weeks of follow-up period.

SUMMARY:
It has been demonstrated by many different researches that for patients to work on their lifestyle modifications, it is important that the patients know their exact blood glucose levels. Unlike the HbA1c which can only be determined at the hospital, improvements in blood glucose levels were detected in both the Type 1 Diabetes Mellitus patients who use insulin as well as Type 2 Diabetes Mellitus patients with SMBG(self-monitoring of blood glucose) which is the method used by patients to measure the blood glucose level at home on their own. Where SMBG needed blood to be collected from the fingertips, it has now passed the continuous glucose monitoring(CGM) stage where blood drawing is no longer required and is now replaced by the real-time CGM(RT-CGM) where blood glucose level can be checked real time. Type 2 Diabetes Mellitus patients who do not use preprandial rapid insulin were divided into SMBG group and intermittent RT-CGM user group and their blood glucose level decrease monitored for 3 months. After 3 months, HbA1c in SMBG group decreased 0.5% compared to the baseline while 1.0% decreased in RT-CGM group. The research was extended 40 weeks to make the total research period to 52 weeks and the results still showed that there were significant decrease in the RT-CGM group. However, up to this day, there are no researches that can show that there are additional decrease in the blood glucose level in Type 2 Diabetes Mellitus patients with use of RT-CGM in the group where sufficient blood glucose management cannot be achieved through use of three oral drug combination therapy to lower the blood glucose level.

This research seeks to find out if there are any decreases in the blood glucose level by using RT-CGM at 6 month period in Type 2 Diabetes Mellitu patient group whose blood glucose level cannot significantly be managed after the three oral hypoglycemic agent combination therapy.

DETAILED DESCRIPTION:
* Pilot, Prospective, open label, multicenter, 3 arm, randomized, feasibility study
* Divided into below three groups iPRo2 only (Control group) / iPRo2 + RT-CGM 1 week treatment (Treatment group 1) / iPRo2 + RT-CGM 1 week on /3 weeks off (2 cycles) (Treatment group 2)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 30 - 65 years old(based on birthdays)
* Type 2 Diabetes Mellitus patients
* Patients who have been taking three types of oral hypoglycemic agent for at least 12 weeks
* Patients whose selection test show HbA1c as 7.5 ~ 10%
* Patients who are willing to use the RT-CGM
* Patients who have signed the letter of consent

Exclusion Criteria:

* Type 1 Diabetes Mellitus patients
* Gestational Diabetes patients
* Patients who have undergone continuous or intermittent insulin treatments for more than 7 days within 12 weeks from the selection test date.
* Patients who underwent oral or non-oral corticosteroid treatment for more than 7 continuous days 1 month before the selection test date.
* Patients with history of hyperplastic diabetic retinosis
* Patients with serious case of infection, scheduled for surgery, history of recent surgery, severe injury
* Patients with history of malignant tumor in five years
* Patients whose records show history of drug abuse or alcoholism within 12 weeks from the questionnaire, medical report and past treatment reports
* Female patients who are pregnant or breast -feeding
* Patients who are participating in other clinical researches other than the current clinical research or who have taken other clinical test drugs within 4 weeks
* Patients who are unfit to partake in this clinical research as determined by the researcher

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c(%) | at 6 month
  This study aimed to see HbA1c(%) changes from baseline and 6month time frame.

SECONDARY OUTCOMES:
the target blood sugar (blood glucose) range | at 6 month
  Comparing indicators such as CGM glycological matrices, Time in Range, etc. at 6 months period to the baseline in each group. Time in range is the amount of time you spend in the target blood sugar (blood glucose) range-between 70 and 180 mg/dL as a normal.
changes in blood pressure(mmHg) | at 6 month
  Comparing the changes in blood pressure to the baseline in each group at 6 month period.
changes in lipid parameter(mg/dl) | at 6 month
  Comparing the changes in lipid parameter to the baseline in each group at 6 month period.
changes in body weight(kg) | at 6 month
  Comparing the changes in body weight to the baseline in each group at 6 month period.
changes in patient satisfaction level | at 6 month
  Comparing the changes in patient satisfaction level to the baseline in each group at 6 month period. (assessed by The Summary of Diabetes Self-Care Activities Measure,

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No